CLINICAL TRIAL: NCT04033874
Title: Comparison of the Efficacy of Non-pharmacological Interventions on Pain Levels, Crying Times and Voice Decibels in Newborns: A Randomized Controlled Trial
Brief Title: The Efficacy of Non-pharmacological Interventions on Pain Levels, Crying Times and Voice Decibels in Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Eskisehir Osmangazi University
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Newborn
Keywords: Heel stick; Newborn; NIPS; Pain levels; Crying times; Voice decibels
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: The prospective, randomized controlled trial including pre and post tests of four groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kangaroo care (Experimental): Heel stick procedure will be performed during kangaroo care.
  During the application, pulse oximetry device will be placed on each newborn right wrist, then heart rate and SpO2 values will be recorded before, during and after the procedure. The device will remain attached to the baby's wrist during the procedure. Then, the pain level will be assessed with NIPS (Neonatal Infant Pain Scale) and heel-stick procedure will be initiated. To determine the crying time, the stopwatch shall be turned on and the sound decibel meter shall be turned on to determine the sound decibel. The general pain level of the newborns will be evaluated by one minute before the procedure and their response to the pain for three minutes during and after the procedure.
  Interventions: Other: kangaroo care
- Mother's lap (Experimental): Heel stick procedure will be performed during newborns who are holding on their mother's lap.
  During the application, pulse oximetry device will be placed on each newborn right wrist, then heart rate and SpO2 values will be recorded before, during and after the procedure. The device will remain attached to the baby's wrist during the procedure. Then, the pain level will be assessed with NIPS (Neonatal Infant Pain Scale) and heel-stick procedure will be initiated. To determine the crying time, the stopwatch shall be turned on and the sound decibel meter shall be turned on to determine the sound decibel. The general pain level of the newborns will be evaluated by one minute before the procedure and their response to the pain for three minutes during and after the procedure.
  Interventions: Other: holding on the mother's lap
- White noise (Experimental): Heel stick procedure will be performed during newborns listened to white noise.
  For the white noise; the track named "do not cry your baby, pt. 2" will be played in Orhan Osman's Colic album. The white noise level will be adjusted to an average of 55 decibels. During the application, pulse oximetry device will be placed on each newborn right wrist, then heart rate and SpO2 values will be recorded before, during and after the procedure. The device will remain attached to the baby's wrist during the procedure. Then, the pain level will be assessed with NIPS (Neonatal Infant Pain Scale) and heel-stick procedure will be initiated. To determine the crying time, the stopwatch shall be turned on and the sound decibel meter shall be turned on to determine the sound decibel. The general pain level of the newborns will be evaluated by one minute before the procedure and their response to the pain for three minutes during and after the procedure.
  Interventions: Other: white noise listening
- Ambient sound (Experimental): Heel stick procedure will be performed during newborns listened to ambient sound.
  During the application, pulse oximetry device will be placed on each newborn right wrist, then heart rate and SpO2 values will be recorded before, during and after the procedure. The device will remain attached to the baby's wrist during the procedure. Then, the pain level will be assessed with NIPS (Neonatal Infant Pain Scale) and heel-stick procedure will be initiated. To determine the crying time, the stopwatch shall be turned on and the sound decibel meter shall be turned on to determine the sound decibel. The general pain level of the newborns will be evaluated by one minute before the procedure and their response to the pain for three minutes during and after the procedure.
  Interventions: Other: ambient sound listening

INTERVENTIONS:
Other: kangaroo care — kangaroo care
  Arms: Kangaroo care
Other: holding on the mother's lap — holding on the mother's lap
  Arms: Mother's lap
Other: white noise listening — white noise listening
  Arms: White noise
Other: ambient sound listening — ambient sound listening
  Arms: Ambient sound

SUMMARY:
This study aimed to investigate and compare the effects of different non-pharmacological interventions (kangaroo care, holding on mother's lap, white noise listening, ambient sound listening) on newborns' crying times, voice decibels and pain levels during heel-stick procedure

DETAILED DESCRIPTION:
The study is a prospective, randomized controlled trial including pre and post tests of four groups. The population of the study consisted of newborns who were followed in the Neonatal Service of Eskişehir City Hospital. The number of newborns to be sampled was determined by power analysis. With a 95% confidence interval, 0.25 effect size and 0.85 strength, 34 newborns are planned to be included in each group. Newborns who meet the inclusion criteria will be randomly assigned to the groups.

In the randomization process; in the four-group design, the rooms were randomly assigned to the study groups by drawing lots in order to eliminate the probability of influence of newborns from each other. Internal blinding was used as a blinding method in order to ensure complete randomization and to prevent Rosental effect. The randomization was performed by the responsible nurse of the unit who was unaware of the pre-test and post-tests of the application.

1. Four different groups were formed in order to prevent the causes of concern in the randomization of patients who were leveled according to their clinical status in the neonatal intensive care unit.
2. In the absence of neonatal intensive care environment noise, four groups were considered due to the limitation in explaining the benefit, contribution and effect of white noise, kangru care and being in the lap of the mother in reducing pain.
3. The newborns treated with kangaroo care and the mother's lap will be the control groups of each other and the newborns treated with white noise and ambient sound will be the control groups of each other.

Research hypotheses:

H1. Newborns receiving kangaroo care during the heel-stick procedure have lower pain levels than newborns who are holding on their mother's lap.

H2. Newborns receiving kangaroo care during the heel-stick procedure have less crying time than newborns who are holding on their mother's lap.

H3. The highest level of sound decibels in the crying process of newborns who receiving kangaroo care during the heel-stick procedure are less than newborns who are holding on their mother's lap.

H4. Newborns listened to white noise during the heel-stick procedure have lower pain levels than newborns who listened to ambient sound.

H5. Newborns listened to white noise during the heel-stick procedure have less crying time than newborns who listened to ambient sound.

H6. The highest level of sound decibels in the crying process of newborns who listened to white noise during the heel-stick procedure are less than newborns listened to ambient sound.

In the study, NIPS (Neonatal Infant Pain Scale) will be used to evaluate the pain severity of newborns in addition to the data form prepared by the researchers.

During the application, pulse oximetry device will be placed on each newborn right wrist, then heart rate and SpO2 values will be recorded before, during and after the procedure. The device will remain attached to the baby's wrist during the procedure. Then, the pain level will be assessed with NIPS and heel-stick procedure will be initiated. To determine the crying time, the stopwatch shall be turned on and the sound decibel meter shall be turned on to determine the sound decibel. The general pain level of the newborns will be evaluated by one minute before the procedure and their response to the pain for three minutes during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Gestation age is between 34-42 weeks
* Birth weight is between 2500-4000 gr
* Apgar score of 1 minute and 5 minutes 8 and above
* Passing the newborn hearing screening test
* To being followed in the neonatal intensive care unit
* To being fed at least half an hour before the procedure
* To being agreed to participate in the study by parents
* To being never received mechanical ventilation / CPAP support after birth
* Having none of congenital anomaly

Exclusion Criteria:

* Inability to take blood the first attempt, as the pain level may change
* Failure of the newborn to pass the hearing screening test
* Newborns hospitalized from polyclinic and emergency department because heel blood was taken before
* Refusing to participate in the study by parents

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Crying times | Five months
  Newborns' crying times during heel-stick procedure will be assessed with the stopwatch
Voice decibels | Five months
  Newborns' voice decibels during heel-stick procedure will be assessed with the sound decibel meter
Pain levels | Five months
  Newborns' pain levels during heel-stick procedure will be assessed with NIPS (Neonatal Infant Pain Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Örsal, Ph.D., Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to share the data of this study in December 2019

REFERENCES:
- [Result] Gao H, Xu G, Gao H, Dong R, Fu H, Wang D, Zhang H, Zhang H. Effect of repeated Kangaroo Mother Care on repeated procedural pain in preterm infants: A randomized controlled trial. Int J Nurs Stud. 2015 Jul;52(7):1157-65. doi: 10.1016/j.ijnurstu.2015.04.006. Epub 2015 Apr 9. PMID 25912524
- [Result] Johnston C, Campbell-Yeo M, Disher T, Benoit B, Fernandes A, Streiner D, Inglis D, Zee R. Skin-to-skin care for procedural pain in neonates. Cochrane Database Syst Rev. 2017 Feb 16;2(2):CD008435. doi: 10.1002/14651858.CD008435.pub3. PMID 28205208
- [Result] Zhu J, Hong-Gu H, Zhou X, Wei H, Gao Y, Ye B, Liu Z, Chan SW. Pain relief effect of breast feeding and music therapy during heel lance for healthy-term neonates in China: a randomized controlled trial. Midwifery. 2015 Mar;31(3):365-72. doi: 10.1016/j.midw.2014.11.001. Epub 2014 Nov 11. PMID 25467598